CLINICAL TRIAL: NCT01050738
Title: Local Analgesia in Knee- and Hipatroplastic Surgery in Patients With Rheumatic Disease: Extra- vs. Intracapsulare Position of Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spenshult Hospital (Other)
Responsible Party: Stefan Bergman/MD, PhD, Research Director, R&D-center Spenshult
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOUS09002
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Rheumatoid Arthritis; Orthopedic Surgery; Analgesia
MeSH Terms: conditions — Arthritis, Rheumatoid; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intracapsulare position (Active Comparator)
  Interventions: Procedure: Position of catheter
- Extracapsulare position (Active Comparator)
  Interventions: Procedure: Position of catheter

INTERVENTIONS:
Procedure: Position of catheter — Position of catheter for administration of local anestesia.

SUMMARY:
Postoperative pain is part of surgery trauma. In orthopedic surgery artroplastic replacement of knee- and hipjoints are common. Postoperative pain relieve can be complicated. A new concept for pain relieve postoperative is local infiltration analgesia (LIA). This technique implicates that a catheter is left in the surgical area and that local anestesia can be administered post surgery. The goal is no or only little pain with minimal side effects. The catheter could be placed intra- or extracapsulare. The best position is not known. Primary aim is to study if position of the catheter effects the need of other postoperative analgesia. Secondary aim is to study if the position effects patient mobility within the first two days.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroplastic surgery of knee or hip

Exclusion Criteria:

* Sensitivity to local anesthetics
* Other reason not to use local anesthetics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Need for other postoperative analgesia. | 48 hours

SECONDARY OUTCOMES:
Patient mobility within the first 48 hours. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bergman, MD, PhD, Study Chair — R&D-center Spenshult
Locations (1):
- Spenshult Hospital, Oskarström, Sweden